CLINICAL TRIAL: NCT03152409
Title: Salicylic Augmentation in Depression
Acronym: SAD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate resources to complete the study
Sponsor: Jessica Harder (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor-Investigator, Jessica Harder, Principle Investigator, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017P000525
Record Dates: First submitted 2017-04-13; First posted 2017-05-15 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Depression; Depressive Disorder; Major Depressive Disorder; Treatment Resistant Depression
Keywords: Aspirin; Treatment; Salicylic acid; anti-inflammatory
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Aspirin; Salicylic Acid

STUDY DESIGN:
Intervention Model Description: Randomized control trial with about half of all participants receiving placebo.
Who Masked: Participant, Investigator
Masking Description: Study team will be blinded to participant condition. Pharmacy will be responsible for providing study drug versus identical placebo to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Aspirin augmentation to treatment (Active Comparator): Participants who meet inclusion criteria for the study and are randomized to the active treatment arm will be given pills for the ensuing 8 weeks, consisting of a daily dose of aspirin 325 mg to be taken every evening before bed.
  Interventions: Drug: Aspirin 325mg
- Placebo augmentation to treatment (Placebo Comparator): Participants randomized to the placebo arm will receive a placebo oral tablet of the same size, shape, and color as the aspirin tablet. Participants will be instructed to take their pills in the evening before bed.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Aspirin 325mg — Participants will take intervention drug dose once a day in combination with their existing antidepressant treatment regimen.
  Other Names: Aspirin; Bayer; Salicylic acid
  Arms: Aspirin augmentation to treatment
Drug: Placebo Oral Tablet — Participants will take a placebo tablet of the same size, shape, and color as the aspirin tablet.
  Other Names: Placebo
  Arms: Placebo augmentation to treatment

SUMMARY:
The investigators are doing this research study to find out if using aspirin along with antidepressant treatment can lessen symptoms of depression. This study also aims to find out if some people improve more from taking aspirin than others. The investigators also want to see if it is possible to predict which participants will do better based on a blood test.

Aspirin is approved by the U.S. Food and Drug Administration (FDA) as an over-the-counter pain medication. But, aspirin is not approved by the FDA to make antidepressant treatment better.

This research study will compare aspirin to placebo.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-control trial. The primary aims of this study are:

Aim 1: To evaluate the clinical effect of aspirin augmentation on depression.

Aim 2: To assess the inflammatory profile of the blood of the aspirin augmentation responders compared with the non-responders.

Aim 3: To evaluate whether immune gene expression patterns are associated with antidepressant response to aspirin.

Aim 4: To collect samples for later, more detailed immunologic characterization.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of major depressive disorder
* Hamilton Depression Rating Scale (HDRS) score of >19
* Stable treatment regimen (no medication changes or changes in psychotherapy treatment in past 8 weeks, and no participation in stepped treatments, such as completion of a course of cognitive behavioral therapy, during the trial)
* Failed to remit with at least 1 antidepressant trial, or combination of 1 antidepressant and 1 augmentation agent
* Women of childbearing age must agree to use an approved method of contraception for the duration of the study

Exclusion Criteria:

* Active suicidal ideation
* History of manic episodes or psychosis
* Alcohol or substance use disorder up to one month prior to first testing session
* Comorbid neurologic condition affecting the central nervous system
* Comorbid autoimmune condition
* Uncorrected thyroid disease or a current abnormal thyroid-stimulating hormone (TSH)
* Active or recent (within the past month) infection (such as otitis, pneumonia, urinary tract infection); temperature > 100.3 or white blood cell (WBC) count > 11 K/microL will be considered evidence of active infection even in the absence of other symptoms
* History of GI bleed
* History of stroke
* History of a bleeding disorder
* Platelet count < 150,000/mm3 on initial screening
* On a blood-thinning agent or taking NSAIDs daily
* Current use of oral steroids or other immunomodulating medications
* Salicylate sensitivity
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Harder, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philip NS, Carpenter LL, Tyrka AR, Price LH. Pharmacologic approaches to treatment resistant depression: a re-examination for the modern era. Expert Opin Pharmacother. 2010 Apr;11(5):709-22. doi: 10.1517/14656561003614781. PMID 20151847
- [Background] Berk M, Dean O, Drexhage H, McNeil JJ, Moylan S, O'Neil A, Davey CG, Sanna L, Maes M. Aspirin: a review of its neurobiological properties and therapeutic potential for mental illness. BMC Med. 2013 Mar 18;11:74. doi: 10.1186/1741-7015-11-74. PMID 23506529
- [Background] Iyengar RL, Gandhi S, Aneja A, Thorpe K, Razzouk L, Greenberg J, Mosovich S, Farkouh ME. NSAIDs are associated with lower depression scores in patients with osteoarthritis. Am J Med. 2013 Nov;126(11):1017.e11-8. doi: 10.1016/j.amjmed.2013.02.037. Epub 2013 Aug 29. PMID 23993259
- [Background] Muller N, Schwarz MJ, Dehning S, Douhe A, Cerovecki A, Goldstein-Muller B, Spellmann I, Hetzel G, Maino K, Kleindienst N, Moller HJ, Arolt V, Riedel M. The cyclooxygenase-2 inhibitor celecoxib has therapeutic effects in major depression: results of a double-blind, randomized, placebo controlled, add-on pilot study to reboxetine. Mol Psychiatry. 2006 Jul;11(7):680-4. doi: 10.1038/sj.mp.4001805. Epub 2006 Feb 21. PMID 16491133
- [Background] Eyre HA, Air T, Proctor S, Rositano S, Baune BT. A critical review of the efficacy of non-steroidal anti-inflammatory drugs in depression. Prog Neuropsychopharmacol Biol Psychiatry. 2015 Mar 3;57:11-6. doi: 10.1016/j.pnpbp.2014.10.003. Epub 2014 Oct 16. PMID 25455584
- [Background] Gallagher PJ, Castro V, Fava M, Weilburg JB, Murphy SN, Gainer VS, Churchill SE, Kohane IS, Iosifescu DV, Smoller JW, Perlis RH. Antidepressant response in patients with major depression exposed to NSAIDs: a pharmacovigilance study. Am J Psychiatry. 2012 Oct;169(10):1065-72. doi: 10.1176/appi.ajp.2012.11091325. PMID 23032386
- [Background] Akhondzadeh S, Jafari S, Raisi F, Nasehi AA, Ghoreishi A, Salehi B, Mohebbi-Rasa S, Raznahan M, Kamalipour A. Clinical trial of adjunctive celecoxib treatment in patients with major depression: a double blind and placebo controlled trial. Depress Anxiety. 2009;26(7):607-11. doi: 10.1002/da.20589. PMID 19496103
- [Background] Abbasi SH, Hosseini F, Modabbernia A, Ashrafi M, Akhondzadeh S. Effect of celecoxib add-on treatment on symptoms and serum IL-6 concentrations in patients with major depressive disorder: randomized double-blind placebo-controlled study. J Affect Disord. 2012 Dec 10;141(2-3):308-14. doi: 10.1016/j.jad.2012.03.033. Epub 2012 Apr 18. PMID 22516310

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After completing informed consent, participants who agreed to participate in the study began study procedures; those with a positive pregnancy test, significant abnormalities in blood counts, electrolytes, kidney function, or thyroid stimulating hormone levels, major psychiatric comorbidities, severe current active suicidality, or certain medical conditions were not eligible to be randomized and were excluded prior to group assignment.
Groups:
- Aspirin Augmentation to Treatment: Daily dose of aspirin 325 mg in combination with their existing antidepressant treatment regimen.
- Placebo Augmentation to Treatment: Daily placebo oral tablet of the same size, shape, and color as the aspirin tablet in combination with their existing antidepressant treatment regimen.
Period: Overall Study
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment
Started | 6 | 5
Completed | 3 | 3
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo Augmentation to Treatment: Daily dose of placebo in combination with their existing antidepressant treatment regimen.
- Total: Total of all reporting groups
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Hamilton Depression Rating Scale (HDRS) Score [Mean (Full Range); unit: units on a scale] — Hamilton Depression Rating Scale measures depression symptoms. The minimum score on this scale is 0. The maximum score on this scale is 52. Higher values correspond with more severe depression symptoms. There are no subscales.
  units on a scale | 20.5 [19 to 24] | 21.4 [20 to 26] | 20.9 [19 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Change in Hamilton Depression Scale Score
Description: Change in HDRS score in the treatment versus control groups.
Time Frame: 8 weeks
Population: Analysis population consisted of study completers for whom HDRS scores from final study visit were available.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment
Number analyzed (Participants) | 4 | 3
units on a scale | -9.75 [-16 to 5] | -11.67 [-21 to -7]

2. Secondary Outcome: Response of Inflammatory Biomarkers
Description: Response of inflammatory biomarkers in treatment responders versus treatment non-responders at 8 weeks.
Time Frame: 2 years
Population: No participant inflammatory data were collected. Although blood samples were collected for planned inflammatory assays, the samples were frozen and assays were never performed. Once study was terminated prematurely (due to lack of resources) no further funds were allocated to the study. Thus inflammatory assays could not be funded and inflammatory data analysis could not proceed.
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Biomarker Association With Antidepressant Response
Description: Ability to observe the degree of biomarker association with antidepressant response.
Time Frame: 2 years
Population: Unable to analyze biomarker association with antidepressant response as there was no biomarker data to analyze (study was terminated due to insufficient resources to continue, and biomarker assays were thus never completed).
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Aspirin Augmentation to Treatment | Placebo Augmentation to Treatment
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/5
Other Adverse Events (participants affected / at risk) | 2/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin Augmentation to Treatment (N=6) | Placebo Augmentation to Treatment (N=5)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Bone fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Symptoms of existing major depression (Psychiatric disorders) | 1 (1) | 2 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aspirin Augmentation to Treatment (N=6) | Placebo Augmentation to Treatment (N=5)
Itchiness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Menstrual symptoms (Reproductive system and breast disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 1
Dental / oral problems (General disorders) | 1 | 2
GI discomfort or distress (Gastrointestinal disorders) | 1 | 1
Upper respiratory tract infection symptoms (Infections and infestations) | 1 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Urinary tract symptoms (Renal and urinary disorders) | 1 | 0
Depression and related symptoms (Psychiatric disorders) | 1 | 2
Muscle aches (General disorders) | 1 | 1
Dizziness (General disorders) | 1 | 0
Rapid heart rate (Cardiac disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
In Mar. 2020 study placed on prolonged pause due to the pandemic. Research activities resumed with limitations later that year. The last study participant was screened in Feb. 2021. However, personnel departure affected study activities, so study was again paused, with plans to resume once adequate personnel were hired. However no additional support was provided. In Dec. 2022, it was decided to terminate the study when it became clear that resources would be insufficient to complete the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT03152409/Prot_SAP_000.pdf